CLINICAL TRIAL: NCT03514680
Title: Evaluating a Clinician Support Algorithm to Enhance Implementation of Evidence-Based Chemotherapy-Induced Peripheral Neuropathy Assessment and Management Recommendations
Brief Title: Clinician Decision Support Algorithm for Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Robert Knoerl, PhD, RN, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-049
Record Dates: First submitted 2018-04-21; First posted 2018-05-02 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Cancer; Chemotherapy-induced Peripheral Neuropathy
Keywords: Cancer Care; Chemotherapy-induced peripheral neuropathy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The study expect to enroll 162 patients, 60 clinicians, and 30 healthy controls for a total of 252.
  81 patients will be recruited in Period 1 (usual care) and a separate 81 will be recruited in Period 2 (algorithm use). The 60 clinicians will be recruited and will participate in Periods I and II. We will use purposive sampling to recruit 30 health controls to match the age and demographic characteristics of the recruited patients. The healthy controls will receive no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period I (No Intervention): -Consented patients will complete electronic versions of the PRO-CTCAE CIPN severity and interference items, 0 - 10 worst CIPN pain numerical rating scale, and QLQ-CIPN20 via tablet prior to their clinician visit at the outpatient oncology center at three consecutive clinic visits: baseline, visit 2, visit 3.
- Period II (Experimental): * Consented patients will complete the same battery of assessments from the usual care period at the baseline, visit 2, and visit 3 time points.
  * Following patient completion of the screening questionnaires, study staff will provide the clinicians with a color-coded summary of the patients' responses to the screening questionnaires and the CIPN assessment and management algorithm
  Interventions: Behavioral: CIPN Assessment and Management Algorithm

INTERVENTIONS:
Behavioral: CIPN Assessment and Management Algorithm — The revised algorithm incorporates evidence-based CIPN assessment and management strategies and standardized CIPN/pain patient-reported outcomes measures. In terms of processes, trained study staff will administer the screening questionnaires (e.g., PRO-CTCAE, 0 - 10 numerical rating scale of worst CIPN pain intensity) to consented patients before their clinician visit (e.g., in the waiting room). Following patient completion of the screening questionnaires, study staff will provide the clinicians with a color-coded summary of the patients' responses to the screening questionnaires and the CIPN assessment and management algorithm. Clinicians may then use the algorithm at their discretion to guide the assessment and management of their patients' CIPN symptoms
  Arms: Period II

SUMMARY:
This research study is evaluating how well a decision support tool works to improve clinicians' use of recommended chemotherapy-induced peripheral neuropathy (CIPN) assessment and management strategies in participants receiving chemotherapy.

DETAILED DESCRIPTION:
This research study will test a new clinician decision support tool for the assessment and management of CIPN. The algorithm is designed to help clinicians make decisions about which strategies to use for the assessment and/or management of CIPN. The investigators need to recruit participants receiving chemotherapy that is known to cause CIPN to determine how well the algorithm works to increase clinicians' use of recommended CIPN assessment and management strategies.

ELIGIBILITY:
Inclusion Criteria for Patients:

* over 18 years of age,
* completed one infusion of neurotoxic chemotherapy for the treatment of cancer
* has at least three more planned clinic visits associated with neurotoxic chemotherapy receipt after the day of consent
* ambulatory,
* signed informed consent,
* willingness to participate in all study activities,
* speaks/reads English,
* receives care from one of the clinicians enrolled in the study.

Exclusion Criteria for Patients:

* prognosis of ≤ two months or
* documented peripheral neuropathy due to other causes (diabetes, alcohol abuse, central nervous system malignancy, vitamin B deficiency, hereditary, nerve compression injury).

Inclusion Criteria for Clinicians:

-if they are a Medical Doctor, Physician Assistant, or Nurse Practitioner and provide care to oncology patients at one of the study sites

Inclusion Criteria for Healthy Controls:

-if they are an adult (18+) who does not have cancer or symptoms of peripheral nerve injury from any cause and speak/read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Clinician Medical Record Abstraction Form | From enrollment until the date of the patient's visit 3 time point, assessed up to approximately 10 weeks.
  Frequency of clinician CIPN assessment and management documentation for each period.

SECONDARY OUTCOMES:
European Organization of Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy Scale (QLQ-CIPN20): Sensory and Motor Subscales | From enrollment until the date of the patient's visit 3 time point, assessed up to approximately 10 weeks.
  Change in QLQ-CIPN20 scores between periods. Subscale total scores are scored from 0 - 100, higher scores represent worse neuropathy symptoms.
Patient-Reported Outcomes National Cancer Institute Common Terminology Criteria for Adverse Events CIPN Severity and Interference Items | From enrollment until the date of the patient's visit 3 time point, assessed up to approximately 10 weeks.
  Reliability and validity testing of measure. The severity and interference items are scored from 0 - 4, with higher scores representing worse neuropathy.
0 - 10 Worst CIPN Numerical Rating Scale | From enrollment until the date of the patient's visit 3 time point, assessed up to approximately 10 weeks.
  Change in 0 - 10 Worst CIPN Numerical Rating Scale score between periods. Scored from 0 - 10, higher scores represent worse pain.
Adapted Acceptability E - Scale | From enrollment to until all patient participants complete both study periods, assessed up to approximately one year.
  Mean score will be calculated to determine clinician-related acceptability and satisfaction with intervention use. Each item is scored from 1 - 5, with higher scores representing greater acceptability and satisfaction.
Feasibility of Algorithm Implementation | From enrollment to until all patient participants complete both study periods, assessed up to approximately one year.
  Mean score to examine feasibility of intervention feasibility. Each item is scored from 1 - 5, with higher scores representing greater feasibility. Will be completed by clinicians only.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knoerl, PhD, RN, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knoerl R, Mazzola E, Mitchell SA, Hong F, Salehi E, McCleary N, Ligibel JA, Reyes K, Berry DL. Measurement properties of brief neuropathy screening items in cancer patients receiving taxanes, platinums, or proteasome inhibitors. J Patient Rep Outcomes. 2021 Sep 26;5(1):101. doi: 10.1186/s41687-021-00377-z. PMID 34568984
- [Derived] Knoerl R, Mazzola E, Hong F, Salehi E, McCleary N, Ligibel J, Reyes K, Berry DL. Exploring the impact of a decision support algorithm to improve clinicians' chemotherapy-induced peripheral neuropathy assessment and management practices: a two-phase, longitudinal study. BMC Cancer. 2021 Mar 6;21(1):236. doi: 10.1186/s12885-021-07965-8. PMID 33676431